CLINICAL TRIAL: NCT05347121
Title: Evaluation of Neck Ultrasound Measurements as a Difficult Airway Signification
Brief Title: Difficult Airway and Ultrasonographic Evaluation
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Elif Ozge Cınar Kose, MD, Kocaeli University
Other Study IDs: ZUSG1
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Difficult Airway

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- difficult airway
  Interventions: Diagnostic Test: difficult airway

INTERVENTIONS:
Diagnostic Test: difficult airway — ultrasonography of airway

SUMMARY:
In this study, it was planned to evaluate the preoperative neck ultrasonography measurements as a predictor of difficult airway in adult patients who will undergo elective surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical condition I-II-III

Exclusion Criteria:

* . Uncooperative patients,
* pregnant women,
* patients who have had head and neck trauma/surgery,
* patients with a known history of difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included American Society of Anesthesiologists (ASA) physical status I-II-III, 120 patients over the age of 18 who would be operated under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
epiglottis-skin thickness | one month
  epiglottis-skin thickness is a marker of difficult airway

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Üniversitesi, Kocaeli, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided